CLINICAL TRIAL: NCT05667506
Title: A Phase Ib/II, Single Arm, Multi-center Study Evaluating the Safety and Efficacy of CNCT19 in Children and Adolescent(Pediatric) Patients With Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia (r/r B-ALL)
Brief Title: A Study of CNCT19 Treatment in Children and Adolescent r/r ALL Patients(Pediatric)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY001103
Record Dates: First submitted 2022-12-05; First posted 2022-12-28 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: CNCT19; Cluster of differentiation antigen 19(CD19); CD19-directed CAR-T cells
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single dose of CNCT19 (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, CNCT19.
  Interventions: Biological: single dose of CNCT19

INTERVENTIONS:
Biological: single dose of CNCT19 — Autologous 2nd generation CD19-directed CAR-T cells, single infusion intravenously.
  Lymphodepletion treatment:
  Drugs:Fludarabine Drugs: Cyclophosphamide

SUMMARY:
This is a multi-center, phase Ib/II trial to evaluate the safety and efficacy of CNCT19 treatment in Children and Adolescent (pediatric) patients with relapsed or refractory B-cell acute lymphoblastic leukemia (r/r B-cell ALL).

DETAILED DESCRIPTION:
This trial is a multi-center, open label, single-arm, phase Ib/II trial to evaluate the safety and efficacy of CNCT19 in Children and Adolescent(aged 3~18 years old) patients (pediatric) with r/r B-cell ALL.

The phase Ib part of the trial is to evaluate the safety, optimal dose of CNCT19, Pharmacokinetics/Pharmacodynamics(PK/PD)and preliminary efficacy in the treatment of Children and Adolescent patients with r/r B-cell ALL.

The phase II part of the trial is to evaluate the efficacy and safety of CNCT19 in in the treatment of Children and Adolescent patients with r/r B-cell ALL.

The study includes screening, pre-treatment (Cell Product manufacture & lymphodepletion), CNCT19 infusion , safety and efficacy follow-up, and survival follow-up. All subjects who have received CNCT19 infusion will be followed for up to 2 years.

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed written informed consent prior to any study procedures (patient and/or parent or legal guardian)
2. Age 3 to 18. Weight ≥10kg
3. Relapsed or refractory acute lymphoblastic leukemia (ALL).
4. Documentation of CD19 tumor expression demonstrated in bone marrow or peripheral blood within 3 months before screening.
5. Bone marrow with ≥ 5% lymphoblasts by morphologic assessment at screening.
6. Karnofsky (age ≥ 16 years) performance status ≥ 70 or Lansky (age < 16 years) performance status ≥ 50 at screening
7. Organ function requirements: All patients must have adequate renal and liver functions

Key Exclusion Criteria:

1. Active Central Nervous System (CNS) involvement by malignancy.
2. Isolated extra-medullary disease relapse.
3. Patients with Burkitt's lymphoma/leukemia, mixed phenotypic acute leukemia and Chronic Myelogenous Leukemia in Blast Crisis
4. History of concomitant genetic syndrome
5. Patients with acute graft-versus-host disease (GVHD) or moderate-to-severe chronic GVHD within 4 weeks before screening.
6. Active systemic autoimmune disease
7. Known infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus (HbsAg positive) or hepatitis C virus (anti-HCV positive).
8. Patients with active infections at screening.
9. Patients who received specified chemotherapy before CNCT19 infusion
10. Radiotherapy before CNCT19 infusion:

    Non-CNS site of radiation completed < 4 weeks prior to CNCT19 Infusion; CNS directed radiation completed < 8 weeks prior to CNCT19 infusion.
11. Donor lymphocyte infusion (DLI) must be stopped > 6 week prior to CNCT19 infusion.
12. Has had treatment with any prior CAR-T therapy.
13. Life expectancy < 3 months.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Overall Remission Rate (ORR) | within 3 months
  ORR is defined as Complete Remission (CR) and Complete Remission with Incomplete Blood Count Recovery (CRi) per NCCN classification, as determined by Independent Review Committee (IRC)

SECONDARY OUTCOMES:
Overall complete Remission Rate (ORR) with minimal residual disease (MRD) negativity as determined by IRC and Investigators | within 3 months
  MRD negativity status as determined using flow cytometry
Overall Remission Rate (ORR) as determined by IRC and Investigators | at the end of month 3
  The Investigators' evaluation results of ORR will be utilized in the sensitivity analysis
Overall Remission Rate (ORR) with minimal residual disease (MRD) negativity as determined by IRC and Investigators | at the end of Month 3
  MRD negativity as determined using flow cytometry
Best overall response (BOR) | up to 2 years
  The proportion of patients who have achieved the best response (CR or CRi) after CNCT19 treatment
Duration of remission (DOR) | to data cutoff date
  DOR is defined as the time between their first complete response per independent review to relapse or any death in the absence of documented relapse
Allogeneic Stem Cell Transplant (Allo-SCT) rate | First infusion date of CNCT19 to data cutoff date(up to 2 years)
  The proportion of patients who have received Allo-SCT after CNCT19 treatment
Relapse Free Survival (RFS) | 2 years
  RFS is defined as the time from the CNCT19 infusion date to the date of disease relapse or death from any cause.
Overall survival (OS) | 2 years
  OS is defined as the time from the CNCT19 Cell Injection infusion to the date of death from any cause
Treatment-Emergent Adverse Events | up to 2 years
  Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAE) and Severity of TEAE
Percentage of Participants Experiencing Clinically Significant Laboratory Abnormalities | From CNCT19 infusion to date of data cutoff (maximum: 2 years)
  Clinically significant laboratory abnormalities were defined as per investigator's discretion
In vivo cellular Pharmacokinetic (PK) profile of CNCT19 | Up to 3 months(BM sample); Up to 2 years(Blood sample)
  To characterize the concentration of CAR-T cell in peripheral blood, bone marrow and cerebral spinal fluid (CSF, if available)by Flow Cytometry and quantitative polymerase chain reaction(qPCR).
Pharmacokinetic (PK)- Cmax of CNCT19 | Up to 2 years
  Maximum detected concentration of CNCT19 in peripheral blood
Pharmacokinetic (PK)- Tmax of CNCT19. | Up to 2 years
  Time to maximum concentration of CNCT19 in peripheral blood
Pharmacokinetic (PK)- AUC of CNCT19. | Up to 2 years
  Area under the concentration (AUC) vs time curve of CNCT19 in peripheral blood
Concentration of Cytokines in Serum | 28 days
  Collected as pharmacodynamic data, including IL-6 at least
Percentage of participants with anti-CNCT19 antibodies in serum | 2 years
  To characterize prevalence and incidence of humoral immunogenicity to CNCT19

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Zhu, M.D, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (9):
- China (9):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science of Technology, Wuhan, Hubei
  - Children's Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affilicated Hospital of Nanchang University, Nanchang, Jiangxi
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No
Currently the investigators have no plan of interim anaylsis, the investigators don't plan to share individual participant data(IPD) during the trial on-going.